CLINICAL TRIAL: NCT04586894
Title: Atteintes Myocardiques, péricardiques et Vasculaires Sous Simple et/ou Double immunothérapie Anti-cancéreuse Anti-PD1, antiPDL1 et Anti-CTLA4
Brief Title: Adverse Myocardial and Vascular Side Effects of Immune Checkpoint Inhibitors
Acronym: AMICI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fédération Française de Cardiologie (Other); BioSerenity (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP191048; 2020-A01502-37 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Cancer; Immune Defect; Cardiovascular Abnormalities
Keywords: Cardiotoxicity; Immune checkpoint inhibitors; Cancer; Myocarditis; Pericarditis; Myositis; Thrombotic events
MeSH Terms: conditions — Neoplasms; Cardiovascular Abnormalities; Cardiotoxicity; Myocarditis; Pericarditis; Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Diagnostic Test: Cardiac MRI; Device: Smart cloth; Other: Biobanking

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Gadolinium-enhanced magnetic resonance imaging of the heart before the first cycle of chemotherapy
Device: Smart cloth — A smart cloth recording cardiac and hemodynamic parameters will be worn by patients during 42 days. Replaced by a holter monitor if the smart cloth is refused or not tolerated by the patient.
Other: Biobanking — Blood samples (plasma, serum, DNA, stem cells, immune cells) taken as part of the study will be stored in a biological sample collection. These samples may be used for further analysis not described in the initial protocol but which may be useful for investigation or in light of advances in scientific knowledge.

SUMMARY:
Our knowledge on cardiovascular side effects of immune checkpoint inhibitors (ICIs) is restricted to this date to observational retrospective data (mainly case series and pharamcovigilance analysis). We aim at assessing the incidence of cardiovascular adverse side effects of ICIs by means of a prospective interventional single centre study using multiple biomarkers.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICIs) are drastically improving cancer prognosis. Cardiovascular adverse side effects of ICIs are though to be rare but may be responsible for ~50% death rates.

Prospective screening for cardiovascular and muscular immune related side effects has not been undertaken independently from the industry.

The aim is to describe the incidence of these side effects by means of serial assessment in patients undergoing ICI therapy for cancer. Biomarkers as ECG, echocardiography, cardiac magnetic resonance imaging and long-term ECG monitoring will be undertaken at inclusion (before ICI therapy is started), and during the first cycle treatments and at 6 months follow-up.

Mean endpoint encompasses cardiovascular and muscular adverse side effects between the 2nd and the 3rd ICI cycle. Secondary endpoints include cardiovascular and muscular adverse side effects at 6 months follow-up, and the incidence of individual side effects.

4 ancillary studies based on patients' blood biobanking are also planned. Their objectives are:

* to assess sensitivity of heart failure biomarkers in predicting cardiovascular events under ICI,
* to assess sensitivity of cytokine biomarkers in predicting cardiovascular events under ICI,
* to bank cells to induce cardiomyocytes from stem cells
* to bank DNA to identify genetic factors related to occurrence of cardiovascular events under ICI

ELIGIBILITY:
Inclusion Criteria:

- prescribed treatment by immune checkpoint inhibitors (ICI) for cancer

Exclusion Criteria:

* previous treatment by any ICI
* any contraindication to cardiac resonance magnetic imaging
* contraindication to gadoteric acid, meglumin or any gadolinium-based contrast agent
* pace maker or automated implantable defibrilator
* pregnancy, breastfeeding
* women of childbearing potential who do not use one of the following methods of birth control: hormonal contraception or intrauterine device or bilateral tubal occlusion
* patient under legal protection
* renal failure defined by creatinine clearance <30ml/min/m² (CKD-EPI)
* current participation or exclusion period of another interventional clinical study

Exclusion Criteria for ancillary studies:

- hemoglobinemia < 9 g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ICI therapy for cancer before the start of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with major cardiovascular advserse drug reactions | 6 weeks
  Incidence of a composite endpoint including myocarditis, pericarditis, acute coronary syndrome, acute heart failure, subclinial cardio-toxicity, high degree conduction abormalities or ventricular sustained arrythmias, cardiovascular death.

SECONDARY OUTCOMES:
Number of patients with major cardiovascular advserse drug reactions | 6 months
  Incidence of a composite endpoint including myocarditis, pericarditis, acute coronary syndrome, acute heart failure, subclinial cardio-toxicity, high degree conduction abormalities or ventricular sustained arrythmias, cardiovascular death.
Number of patients with other cardiovascular advserse drug reactions | 6 weeks and 6 months
  Incidence of a composite endpoint including vasculitis or myositis.
Number of patients with isolated CMR abnormalities | 6 weeks and 6 months
  Serial assessment
Number of patients with rhythm abnormalities that do not fullfill major advsere event criteria | 6 weeks and 6 months
  Burden of extrasystole, low degree conduction disorders
Risk factors for cardiovascular adverse drug event | 6 weeks and 6 months
  Characterization of risk predictors for occurrence of cardiovascular adverse drug event, among the following: socio-demographic characteristics, oncologic characteristics, previous treatments, serum biomarkers, patient assessment on ESC-SCORE and ACC/AHA ASCVD risk scoring systems, immune status, cardiac characteristics on imaging.

OTHER OUTCOMES:
Biomarkers level of heart failure | Baseline
Cytokinic biomarkers level | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Mirabel, MD, Principal Investigator — Inserm U970 Paris Cardiovascular Research Center
Locations (1):
- AP-HP - Hôpital européen Georges-Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement. Processing of shared data must comply with European General Data Protection Regulation (GDPR).